CLINICAL TRIAL: NCT01235741
Title: A Randomized, Double-Blind, Placebo-Controled, Multicenter Study To Examine The Efficacy And Safety Of Pramlintide+Metreleptin In Obese Subjects Following A Low-Calorie Diet Lead-In
Brief Title: A Study To Examine The Efficacy And Safety Of Pramlintide+Metreleptin In Obese Subjects
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Results from previous study DFA102 demonstrated neutralizing activity to metreleptin in invitro assay in 2 participants.
Sponsor: AstraZeneca (Industry)
Collaborators: Takeda Pharmaceuticals North America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DFA104
Record Dates: First submitted 2010-11-02; First posted 2010-11-08 (Estimated); Results first posted 2013-12-09 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-03

CONDITIONS: Obesity
Keywords: Pramlintide; Metreleptin; Obesity; Amylin; Takeda
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental): Pramlintide+Metreleptin
  Interventions: Drug: Pramlintide+Metreleptin
- Group B (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pramlintide+Metreleptin — Group A: Subcutaneous Injection once a day (QD): Pramlintide 360 mcg+Metreleptin 5.0 mg for 1 week followed by Pramlintide 360 mcg+Metreleptin 5.0 mg twice a day (BID) for 15 weeks.
  Arms: Group A
Drug: Placebo — Group B: Subcutaneous Injection-twice a day (BID): Placebo equivalent volumes to active doses.
  Arms: Group B

SUMMARY:
Following screening, eligible subjects will be enrolled into a 6-week Low Calorie Diet (LCD) lead-in period. Subjects who lose at least 2% of their body weight at the end of the 6-week LCD lead-in period will be randomized to 1 of 2 treatment arms (pramlintide+metreleptin or placebo) to begin a 16-week treatment period during which the effect on body weight of treatment with pramlintide+metreleptin will be compared to placebo. Following the 16 week blinded core treatment period, subjects will discontinue study medication for a period of 12 weeks. Following the 12 week off-drug follow-up period, subjects in both groups will initiate a 12 week open-label treatment period with Pramlintide+Metreleptin. During the 12 week off-drug and 12 week open label treatment periods, subjects will continue to participate in a Lifestyle Intervention (LSI) program.

ELIGIBILITY:
Inclusion Criteria:

* Is obese with a BMI ≥35 to ≤45 kg/m2.
* Has stable body weight (not varying by >5% within 3 months prior to study start).
* Meets certain requirements with respect to concomitant medications.
* Has not smoked or used nicotine-containing products for at least 12 months prior to study start.

Exclusion Criteria:

* Has not been enrolled in a weight loss program within 2 months prior to study start.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 213 (Actual)
Dates: Start 2011-01; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Senior Vice President, Research & Development, Study Director — Amylin Pharmaceuticals, LLC.
Locations (18):
- United States (18):
  - Research Site, Greenbrae, California
  - Research Site, La Jolla, California
  - Research Site, Denver, Colorado
  - Research Site, Winter Park, Florida
  - Research Site, Chicago, Illinois
  - Research Site, Baton Rouge, Louisiana
  - Research Site, Hyattsville, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, St Louis, Missouri
  - Research Site, Butte, Montana
  - Research Site, New York, New York
  - Research Site, Tulsa, Oklahoma
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Austin, Texas
  - Research Site, Salt Lake City, Utah
  - Research Site, Arlington, Virginia
  - Research Site, Norfolk, Virginia
  - Research Site, Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 5 January 2011 Lead-In Period started. 28 September 2011 last participants final visit procedure. Clinics where participants with body mass index [BMI] greater than, equal to (≥)35 kilogram per meter squared (kg/m^2) and less than, equal to (≤)45 kg/m2) could be enrolled.
Pre-assignment Details: 6 week lead-in period:low-calorie diet (LCD); 16 week randomized treatment period: participants who lost >=2% body weight at end of LCD were randomized to an arm. Sponsor terminated study during randomization period due to neutralizing activity to metreleptin observed in Study DFA102, NCT00673387. Safety follow-up 2, 4, 6 months post treatment.
Groups:
- Low Calorie Diet Only: 6 Week Lead-in Period with low calorie diet (LCD); in the last week of the 6 week LCD, self administered subcutaneous (SC) injections of placebo once a day (QD) was initiated and then followed by randomization to either study drug or placebo in the Randomization period.
- Placebo: Self administered subcutaneous (SC) injection of placebo matched to pramlintide (Placebo-P) plus placebo matched to metreleptin (Placebo-M) twice a day (BID) for 16 weeks.
- Pramlintide + Metreleptin: Self administered SC injection of pramlintide 360 micrograms (µg) + metreleptin 5.0 milligrams (mg) BID for 16 weeks
Period: Non-Randomized Low Calorie Diet Lead-In
Arm/Group | Low Calorie Diet Only | Placebo | Pramlintide + Metreleptin
Started | 213 (6 Week LCD period. Those who lost >=2% of body weight were randomized to treatment.) | 0 | 0
Completed | 72 (Study terminated by Sponsor. 72 randomized to treatment at time study halted.) | 0 | 0
Not Completed | 141 | 0 | 0
Not completed — Withdrawal by Subject | 9 | 0 | 0
Not completed — Sponsor terminated study | 121 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Lost to Follow-up | 5 | 0 | 0
Not completed — Failed to meet weight loss in Period 1 | 4 | 0 | 0
Period: Randomized to Treatment
Arm/Group | Low Calorie Diet Only | Placebo | Pramlintide + Metreleptin
Started | 0 | 36 | 36
Completed | 0 | 0 (Study terminated by Sponsor. Maximum exposure to study drug was 30 days.) | 0 (Study terminated by Sponsor. Maximum exposure to study drug was 30 days.)
Not Completed | 0 | 36 | 36
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Adverse Event | 0 | 1 | 1
Not completed — Sponsor terminated study | 0 | 35 | 34
Period: Follow-Up Post Treatment up to Month 6
Arm/Group | Low Calorie Diet Only | Placebo | Pramlintide + Metreleptin
Started | 0 | 36 (No treatment; those who had been treated with placebo (36) were followed up 6 Months post treatment.) | 36 (No treatment; those who had been treated with drug (36) were followed up 6 months post treatment.)
Completed | 0 | 27 (9 participants did not complete the 6 month follow up period) | 29 (7 participants did not complete the 6 month follow up period)
Not Completed | 0 | 9 | 7
Not completed — Withdrawal by Subject | 0 | 3 | 6
Not completed — Lost to Follow-up | 0 | 5 | 1
Not completed — Other | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Baseline for all participants (213) was baseline at enrollment (Day 1 of Lead-in period); baseline for participants who were randomized to treatment before study was terminated was Day 1 of randomization (last measurement before first dose of assigned drug).
Groups:
- Non-Randomized Lead-in LCD: 6 Week Lead-in with low calorie diet (LCD); in the last week of the 6 week LCD, self administered subcutaneous (SC) injections of placebo once a day (QD) was initiated and then followed by randomization to study drug in the Randomization period.
- Placebo: Self administered subcutaneous (SC ) injection of placebo matched to pramlintide (Placebo-P) plus placebo matched to metreleptin (Placebo-M) twice a day (BID) for 16 weeks.
- Pramlintide + Metreleptin: Self administered SC injection of pramlintide 360 µg + metreleptin 5.0 mg BID for 16 weeks
- Total: Total of all reporting groups
Arm/Group | Non-Randomized Lead-in LCD | Placebo | Pramlintide + Metreleptin | Total
Number analyzed (Participants) | 141 | 36 | 36 | 213
Age, Continuous [Mean (Standard Deviation); unit: years] — Age at Screening is presented.
  years | 46.1 (11.81) | 46.2 (10.84) | 46.4 (10.45) | 46.1 (11.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 106 | 27 | 29 | 162
  Male | 35 | 9 | 7 | 51
Region of Enrollment [Number; unit: participants]
  United States | 141 | 36 | 36 | 213
Body Weight [Mean (Standard Deviation); unit: kg] — Body weight at enrollment measured in kilograms (kg).
  kg | 110.86 (13.210) | 109.10 (16.850) | 108.34 (12.032) | 110.13 (13.678)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index (BMI) at enrollment measured in kilograms per meter of height squared (kg/m^2).
  kg/m^2 | 39.51 (2.875) | 39.17 (3.279) | 39.09 (2.869) | 39.38 (2.937)

OUTCOME MEASURES:

1. Secondary Outcome: Percent Change From Baseline to Week 1 and From Baseline to Month 6 Follow-up in Body Weight - Intent to Treat Population
Description: Baseline was Day 1 measurement or the last measurement taken prior to first dose of randomized study medication, if Day 1 measure was missing. Follow up was 6 months post last dose of randomized study medication.
Time Frame: Baseline up to Month 6 Follow-Up
Population: The intent to treat (ITT) population received at least one dose of randomized study treatment. The number analyzed in the ITT included those participants who provided a measurement. Number analyzed (n) for Week 1 provided above; 6 Month Follow-Up n=27, 29, in placebo and Pramlintide + Metreleptin, respectively.
Measure: Mean (Standard Deviation); unit: percentage of change in weight
Groups:
- Placebo: Self administered SC injection of placebo matched to pramlintide (Placebo-P) plus placebo matched to metreleptin (Placebo-M) BID for 16 weeks.
Arm/Group | Placebo | Pramlintide + Metreleptin
Number analyzed (Participants) | 20 | 23
percentage of change in weight
  Week 1 | -0.34 (0.924) | -0.26 (0.819)
  6 Month Follow-Up | -0.02 (6.575) | -1.80 (6.063)

2. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events and Number With Post Treatment Adverse Events - Intent to Treat Population
Description: Treatment-Emergent Adverse Events are defined as those with an onset date and time on or after the first dose of randomized study medication and on or before the last dose of randomized study medication. Post-treatment Adverse Events are defined as those with an onset date after the date of last dose (imputed if not available) of randomized study medication. Participants experiencing multiple episodes of a given adverse event are counted once.
Time Frame: Day 1 up to Month 6 Follow-Up
Population: The intent to treat (ITT) population received at least one dose of randomized study treatment.
Measure: Number; unit: participants
Groups:
- On Treatment Placebo: Self administered SC injection of placebo matched to pramlintide (Placebo-P) plus placebo matched to metreleptin (Placebo-M) BID for 16 weeks.
- On Treatment Pramlintide + Metreleptin: Self administered SC injection of pramlintide 360 µg + metreleptin 5.0 mg BID for 16 weeks
- Post Treatment Placebo Arm; Post Treatment Pramlintide + Metreleptin Arm: From date after the date of last dose (imputed if not available) of randomized study medication up to 6 Months post treatment.
Arm/Group | On Treatment Placebo | On Treatment Pramlintide + Metreleptin | Post Treatment Placebo Arm | Post Treatment Pramlintide + Metreleptin Arm
Number analyzed (Participants) | 36 | 36 | 36 | 36
participants | 6 | 13 | 13 | 16

3. Primary Outcome: Change From Baseline to Week 2, and to Follow up Months 2, 4, 6 in Fasting Leptin Concentration - Intent to Treat Population
Description: Participants who received metreleptin were analyzed; no placebo treated participants were analyzed. Baseline was Day 1 measurement or the last measurement taken prior to first dose of randomized study medication, if Day 1 measure was missing. Leptin was measured in nanograms per milliliter (ng/mL).
Time Frame: Baseline to Month 6 Follow Up
Population: All participants who received a dose of metreleptin and provided a sample were analyzed. Number of participants analyzed for Week 2, and follow up Months 2, 4, 6 were 6, and 33, 29, 29, respectively.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Pramlintide + Metreleptin
Number analyzed (Participants) | 36
ng/mL
  Change from baseline to Week 2 of treatment | 223.38 (512.088)
  Change from baseline to Month 2 Follow up | 15.46 (34.885)
  Change from baseline to Month 4 Follow up | 20.08 (35.732)
  Month 6 Follow up | 10.70 (18.913)

4. Primary Outcome: Number of Participants With Anti-leptin Antibodies Who Received Metreleptin - Intent to Treat Population
Description: Anti-leptin antibodies measured at Weeks 1 and 2 of drug treatment, early termination visit, and at Months 2, 4, and 6 post treatment follow-up in participants who received metreleptin.
Time Frame: Week 1 to Month 6 Follow-Up
Population: All participants who received at least one dose of metreleptin and provided a sample to analyze; number analyzed (n) for Week 1, Week 2, early termination, Month 2, Month 4, Month 6 Follow-up were: n=22, 5, 35, 32, 25, 28.
Measure: Number; unit: participants
Arm/Group | Pramlintide + Metreleptin
Number analyzed (Participants) | 36
participants
  Week 1 | 0
  Week 2 | 1
  Early Termination | 9
  Month 2 Follow-Up | 15
  Month 4 Follow-Up | 10
  Month 6 Follow-Up | 8

5. Primary Outcome: Number of Participants With Neutralizing Activity to Metreleptin at Early Termination or During Post Treatment Follow-Up - Intent to Treat Population Who Received Metreleptin
Description: In vitro assays were conducted to determine if neutralizing activity to metreleptin developed in participants treated with at least one dose of the drug during the study. Baseline is Day 1 of the Randomization Period, prior to administration of metreleptin.
Time Frame: Baseline to Month 6 Follow-Up
Measure: Number; unit: participants
Arm/Group | Pramlintide + Metreleptin
Number analyzed (Participants) | 36
participants | 0

6. Primary Outcome: Number of Participants With Hematology and Urinalysis Laboratory Values of Potential Clinical Importance - Intent to Treat Population
Description: Criteria for laboratory values of potential clinical importance for obese and overweight (BMI >= 25 kg/m^2) participants: Platelets high (H) >500,000/µL; low (L) <75,000/µL. Hematocrit males <36%, females <30%. Hemoglobin males <12 g/dL, females <10 g/dL. White blood cell count (WBC) H >18,000/µL; L <1,500/µL. Urine protein H >= 3+ or >= 500 mg/dL. Urine glucose H >= 3+ or >= 500 mg/dL. Urine ketones >= 3+ or Large.
Time Frame: Screening to 6 Month Follow-Up
Population: The intent to treat (ITT) population received at least one dose of randomized study treatment. Number analyzed (n) in ITT included participants who provided a laboratory measurement. Hemoglobin, hematocrit n=27, 29 in placebo and pramlintide + metreleptin, respectively; urinalysis n=31, 29, in placebo and pramlintide + metreleptin, respectively.
Measure: Number; unit: participants
Arm/Group | Placebo | Pramlintide + Metreleptin
Number analyzed (Participants) | 36 | 36
participants
  Hematocrit | 0 | 1
  Hemoglobin | 0 | 1
  Glucose in Urine | 0 | 1

7. Primary Outcome: Number of Participants With Chemistry Laboratory Value of Potential Clinical Importance - Intent to Treat Population
Description: Criteria for laboratory values of potential clinical importance for obese and overweight (BMI >= 25 kg/m^2) participants: Total bilirubin High (H) > 2 mg/dL; Plasma or serum glucose fasting or non-fasting H > 200 mg/dL, low (L) < 60 mg/dL; Albumin L <2.5 g/dL; Creatine kinase H > 3*Upper limit of Normal (ULN); Sodium L <130 milliequivalents per liter (mEq/L), H > 150 mEq/L; potassium L<3.0 mEq/L, H> 5.5 mEq/L; bicarbonate L<18 mEq/L, H>35 mEq/L;calcium L <8mg/dL, H> 11 mg/dL; triglycerides H> 500 mg/dL; Cholesterol L < 100 mg/dL, H > 350 mg/dL; Alkaline phosphatase H > 3*ULN; Gamma-glutamyltransferase H>3*ULN; creatinine males > 1.6 mg/dL, females > 1.4 mg/dL; alanine aminotransferase H > 3*ULN; aspartate aminotransferase H > 3*ULN; urea nitrogen H > 45 mg/dL; uric acid males > 10.0 mg/dL, females > 8.0 mg/dL; Phosphorus L < 1.0 mg/dL H > 6.0 mg/dL.
Time Frame: Screening to Month 6 Follow-Up
Population: The intent to treat (ITT) population received at least one dose of randomized study treatment. The number analyzed in the ITT included those participants who provided a laboratory measurement.
Measure: Number; unit: participants
Arm/Group | Placebo | Pramlintide + Metreleptin
Number analyzed (Participants) | 36 | 36
participants
  Creatine Kinase | 2 | 3
  Urate | 0 | 2
  Bilirubin | 0 | 1

8. Primary Outcome: Mean Change From Baseline to Month 6 Follow-Up in Blood Pressure - Intent to Treat Population
Description: Baseline was Day 1 measurement or the last measurement taken prior to first dose of randomized study medication, if Day 1 measure was missing. Follow-up was up to 6 months post treatment. Blood pressure included systolic and diastolic pressures measured in millimeters of mercury (mmHg).
Time Frame: Baseline to Month 6 Follow-Up
Population: The intent to treat (ITT) population received at least one dose of drug treatment. The number analyzed in the ITT included those participants who provided a vital sign measurement up to 6 Months follow-up.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Placebo | Pramlintide + Metreleptin
Number analyzed (Participants) | 27 | 29
mmHg
  Systolic Blood Pressure | 4.3 (9.40) | 3.1 (8.90)
  Diastolic Blood Pressure | 2.7 (7.40) | 2.7 (8.07)

9. Primary Outcome: Mean Change From Baseline to Month 6 Follow-Up in Heart Rate - Intent to Treat Population
Description: Baseline was Day 1 measurement or the last measurement taken prior to first dose of randomized study medication, if Day 1 measure was missing. Heart rate was measured in beats per minute (beats/min).
Time Frame: Baseline up to Month 6 Follow-Up
Population: The intent to treat (ITT) population received at least one dose of randomized study treatment. The number analyzed in the ITT included those participants who provided a vital sign measurement.
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | Placebo | Pramlintide + Metreleptin
Number analyzed (Participants) | 27 | 29
beats/min | 1.2 (8.85) | 1.2 (7.98)

10. Primary Outcome: Mean Change From Baseline to 6 Month Follow-Up in Fasting Plasma Glucose - Intent to Treat Population
Description: Baseline was Day 1 measurement or the last measurement taken prior to first dose of randomized study medication, if Day 1 measure was missing. Follow up was 6 months post last dose of randomized study medication. Fasting glucose measured in milligrams per deciliter (mg/dL).
Time Frame: Baseline to 6 Month Follow-Up
Population: The intent to treat (ITT) population received at least one dose of randomized study treatment. The number analyzed in the ITT included those participants who provided a laboratory measurement up to Month 6 Follow-Up.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Pramlintide + Metreleptin
Number analyzed (Participants) | 25 | 29
mg/dL | 6.8 (8.31) | -1.0 (9.03)

11. Primary Outcome: Mean Change From Baseline to Month 6 Follow-Up in Insulin - Intent to Treat Population
Description: Baseline was Day 1 measurement or the last measurement taken prior to first dose of randomized study medication, if Day 1 measure was missing. Follow up was 6 months post last dose of randomized study medication. Insulin measured in milliunits per liter (mU/L).
Time Frame: Baseline up to Month 6 Follow-Up
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: mU/L
Arm/Group | Placebo | Pramlintide + Metreleptin
Number analyzed (Participants) | 27 | 29
mU/L | 3.41 (8.990) | 3.46 (7.617)

12. Primary Outcome: Mean Change From Baseline to Month 6 Follow-Up in Lipids - Intent to Treat Population
Description: Baseline was Day 1 measurement or the last measurement taken prior to first dose of randomized study medication, if Day 1 measure was missing. Follow up was 6 months post last dose of randomized study medication. Lipids measured included total cholesterol, high density lipoprotein (HDL) cholesterol, low density lipoprotein (LDL) cholesterol, and triglycerides. Lipids were measured in milligrams per deciliter (mg/dL).
Time Frame: Baseline up to Month 6 Follow-Up
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | Pramlintide + Metreleptin
Number analyzed (Participants) | 27 | 29
mg/dL
  Total Cholesterol | 21.7 (19.21) | 14.7 (25.51)
  HDL cholesterol | 7.7 (7.25) | 6.6 (7.60)
  LDL cholesterol | 14.0 (17.47) | 9.6 (21.05)
  Triglycerides | 10.4 (35.12) | 3.0 (38.30)

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse events (AEs) and Serious AEs (SAEs): onset date/ time on or after first dose of randomized study medication and on or before the last dose of randomized study medication.
Description: AE=any new unfavorable symptom, sign, or disease or worsening of a preexisting condition. SAE=medical event that results in death, persistent or significant disability/incapacity, or drug dependency/abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization.
Groups:
- Placebo-P + Placebo-M: Self administered subcutaneous injection once a day (QD) of placebo matched to pramlintide (Placebo-P) plus placebo matched to metreleptin (Placebo-M) for 1 week followed by BID dosing for 15 weeks (16 weeks total).
- Pramlintide + Metreleptin: Self administered subcutaneous injection once a day (QD) of pramlintide 360 micrograms (µg) plus metreleptin 5.0 milligrams (mg ) for 1 week followed by twice a week (BID) dosing for 15 weeks (Total of 16 Weeks treatment).
Arm/Group | Placebo-P + Placebo-M | Pramlintide + Metreleptin
Serious Adverse Events (participants affected / at risk) | 0/36 | 1/36
Other Adverse Events (participants affected / at risk) | 1/36 | 14/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo-P + Placebo-M (N=36) | Pramlintide + Metreleptin (N=36)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo-P + Placebo-M (N=36) | Pramlintide + Metreleptin (N=36)
Nausea (Gastrointestinal disorders) | 1 (1) | 7 (9)
injection site hematoma (General disorders) | 0 (0) | 3 (3)
injection site induration (General disorders) | 0 (0) | 2 (2)
injection site pruritus (General disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.